CLINICAL TRIAL: NCT03798795
Title: Development of an MRI-based Radiomic Model for Non-invasive Tumor Grading of Soft Tissue Sarcomas.
Brief Title: Radiomics for Tumor Grading of Soft Tissue Sarcomas.
Status: Completed | Type: Observational
Sponsor: Technical University of Munich (Other)
Collaborators: University of Washington (Other)
Responsible Party: Sponsor
Other Study IDs: Sarcoma_Grading_Radiomics
Record Dates: First submitted 2019-01-07; First posted 2019-01-10 (Actual); Last update posted 2019-04-10 (Actual); Status verified 2019-04

CONDITIONS: Sarcoma, Soft Tissue
MeSH Terms: conditions — Sarcoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Radiomics is defined as a quantitative high-throughput analysis of imaging data combined with model development aiming to predict biological correlates or clinical endpoints. The investigators of this study hypothesize that radiomic features may correlate with pathology-defined tumor grading in soft tissue sarcoma patients. The aim of this study is to develop a predictive radiomics model for tumor grading determination.

DETAILED DESCRIPTION:
Soft tissue sarcomas (STS) constitute an overall rare malignant entity comprising 1% of all cancers with a yearly incidence rate of 3.8 per 100.000 inhabitants. Therapy decisions are made using clinical and pathological determinants defined by the American Joint Committee on Cancer (AJCC). It involves the TNM staging system that classifies STS by their tumor size (measured as maximal diameter), pathological tumor grading defined by the French Fédération Nationale des Centres de Lutte Contre le Cancer (FNCLCC) and the occurrence of nodal or distant metastases.

For the guidance of therapy, the most important factor constitutes tumor grading. In "low-grade" sarcomas (G1), surgical resection is often sufficient for durable tumor control. In "high risk" STS, however, resection of the tumor is combined with radiotherapy improving locoregional control and eventually survival.

Currently, invasive biopsies followed by pathological work-up are necessary to determine tumor grading. However, bioptic specimens are always restricted to small tumor subvolume.

Medical imaging-based analyses constitutes an alternative tool to characterize tissue. Recent developments in quantitative image analysis and data science have led to the evolvement of "Radiomics". It is defined as an algorithm-based large-scale quantitative analysis of imaging features. It should be considered as a two-step process with (1) extraction of relevant imaging features, and (2) incorporating these features into a mathematical model to ultimately predict patient or tumor-specific outcomes. In previous scientific studies, radiomic models have been associated with survival, tumor progression, and molecular changes including genetic mutations or expression profiles as shown in multiple malignant entities. In addition, radiomic models were able to predict tumor grading e.g. for gliomas, meningiomas, hepatocellular carcinoma or pancreatic neuroendocrine tumors. In contrast to pathology, quantitative image analysis (radiomics) has the principal advantage of analyzing the whole tumor.

In this study, the investigators are aiming to correlate radiomic features with tumor grading of STS. The ultimate goal is to develop a prediction model to non-invasively classify tumor grading. In a first step, the focus will be laid on differentiating "low-grade" and "high-grade" STS. In a second step, "high-grade" STS will be divided into G2 and G3 tumors.

To this end, the investigators will retrospectively analyze a patient cohort of 138 patients (139 tumors) with known tumor grading and available pre-therapeutic MRI-scans. As secondary endpoint overall survival will be determined for all patients. An independent patient cohort from the University of Washington (139 patients) will be used for external validation of the developed models.

ELIGIBILITY:
Inclusion Criteria:

* Histologically proven soft tissue sarcoma
* Available pre-therapeutic MRI with a contrast-enhanced T1 weight fat saturated sequence +/- fat saturated T2 sequences (e.g. STIR)

Exclusion Criteria:

* Indeterminate tumor grading
* Osteosarcoma
* Ewing Sarcoma
* Endoprothesis-dependent MRI artifacts
* Previous radiotherapy or chemotherapy
* Lack of a contrast-enhanced T1 weight fat saturated MRI sequence

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with histologically proven soft tissue sarcomas with known FNCLCC tumor grading determined by biopsy prior to therapy.
Sampling Method: Non-Probability Sample
Enrollment: 285 (Actual)
Dates: Start 2017-10-01 (Actual); Primary Completion 2018-03-31 (Actual); Study Completion 2019-03-01 (Actual)

PRIMARY OUTCOMES:
Pathological tumor grading | Baseline
  Defined by the French Fédération Nationale des Centres de Lutte Contre le Cancer (FNCLCC)

SECONDARY OUTCOMES:
Overall Survival | From initial pathologic diagnosis to the time point of death or the time point of censoring up to 100 months.
  Overall Survival

CONTACTS AND LOCATIONS:
Overall Officials: Stephanie E Combs, MD, Principal Investigator — Technical University of Munich
Locations (1):
- Klinik für RadioOnkologie Strahlentherapie, Munich, Bavaria, Germany

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Liang W, Yang P, Huang R, Xu L, Wang J, Liu W, Zhang L, Wan D, Huang Q, Lu Y, Kuang Y, Niu T. A Combined Nomogram Model to Preoperatively Predict Histologic Grade in Pancreatic Neuroendocrine Tumors. Clin Cancer Res. 2019 Jan 15;25(2):584-594. doi: 10.1158/1078-0432.CCR-18-1305. Epub 2018 Nov 5. PMID 30397175
- [Background] Aerts HJ, Velazquez ER, Leijenaar RT, Parmar C, Grossmann P, Carvalho S, Bussink J, Monshouwer R, Haibe-Kains B, Rietveld D, Hoebers F, Rietbergen MM, Leemans CR, Dekker A, Quackenbush J, Gillies RJ, Lambin P. Decoding tumour phenotype by noninvasive imaging using a quantitative radiomics approach. Nat Commun. 2014 Jun 3;5:4006. doi: 10.1038/ncomms5006. PMID 24892406
- [Derived] Peeken JC, Spraker MB, Knebel C, Dapper H, Pfeiffer D, Devecka M, Thamer A, Shouman MA, Ott A, von Eisenhart-Rothe R, Nusslin F, Mayr NA, Nyflot MJ, Combs SE. Tumor grading of soft tissue sarcomas using MRI-based radiomics. EBioMedicine. 2019 Oct;48:332-340. doi: 10.1016/j.ebiom.2019.08.059. Epub 2019 Sep 12. PMID 31522983